CLINICAL TRIAL: NCT01414348
Title: Managing the Dysexecutive Syndrome Following Traumatic Brain Injury: An Ecologically Valid Rehabilitation Approach
Brief Title: Managing Dysexecutive Syndrome (DS): CIHR 2011-2014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Deirdre Dawson, Dr. Deirdre Dawson, Senior Scientist Rotman Research Institute, Baycrest
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: REB1120
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Traumatic Brain Injury; Cerebrovascular Accident (CVA); Acquired Brain Injury
Keywords: participation; activities of daily living; brain injuries; executive function
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional rehabilitation (Active Comparator): In-home work on problems in daily living.
  Interventions: Behavioral: Conventional rehabilitation.
- Novel rehabilitation approach (Experimental)
  Interventions: Behavioral: Novel rehabilitation approach

INTERVENTIONS:
Behavioral: Conventional rehabilitation. — 1 hour / 2x / week for up to 15 sessions
  Arms: Conventional rehabilitation
Behavioral: Novel rehabilitation approach — 1 hr, 2x/week for up to 15 sessions
  Arms: Novel rehabilitation approach

SUMMARY:
Successful community participation following acquired brain injury (ABI) continues to be an elusive goal for patients, clinicians and researchers. Our pilot work shows that community dwelling survivors of ABI can significantly improve performance on self-identified real- world performance problems and that they can transfer this learning to improve goals not trained in the treatment sessions. We will compare two types of rehabilitation intervention using a randomized controlled trial. We will also interview survivors, their significant others and clinicians regarding their experiences with each intervention to help us discover what works best.

DETAILED DESCRIPTION:
Executive dysfunction is endemic after severe acquired brain injuries (ABIs) and is highly associated with long-lasting psychosocial distress, problems in a multiplicity of everyday activities and overall reduced quality of life. There is increasing evidence to suggest that a novel behavioral intervention is a treatment of choice for executive dysfunction. However few studies have addressed ecological relevance: failing to take into account the significant impact of the complex settings of real life on executive function. More data are desperately needed in this area given the devastating consequences of ABI. We propose to investigate the benefits of two community- based interventions.

ELIGIBILITY:
Inclusion Criteria:

* fluent in written and spoken English,
* have sustained (1) a moderate to severe TBI as defined by a 6-hour GCS of 12 or less OR (2) complicated mild TBI with GCS 13-15 and associated abnormal findings on CT or MRI scan OR (3) other form of acquired brain injury (ABI) that is not related to a congenital, developmental or degenerative disorder but which occurred through a medical problem or disease process including stroke,

Exclusion Criteria: other significant neurological or psychiatric history such as multiple sclerosis or psychiatric illness requiring hospitalization, concurrent moderate to severe depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in performance on COPM | pre, post, 3 month follow-up
  Canadian Occupational Performance Measure: standardized interview

SECONDARY OUTCOMES:
DEX, IADL profile | pre, post, 3 month follow-up
  Perceived and observed impact of dysexecutive syndrome in everyday life

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre D Dawson, PhD, Principal Investigator — Baycrest centre
Locations (1):
- Baycrest Centre for Geriatric Care, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dawson DR, Anderson ND, Binns MA, Bottari C, Damianakis T, Hunt A, Polatajko HJ, Zwarenstein M. Managing executive dysfunction following acquired brain injury and stroke using an ecologically valid rehabilitation approach: a study protocol for a randomized, controlled trial. Trials. 2013 Sep 22;14:306. doi: 10.1186/1745-6215-14-306. PMID 24053695